CLINICAL TRIAL: NCT00157196
Title: A Multi-center, Non-randomized, Open Label Safety Study of BLP25 Liposome Vaccine (L-BLP25) in Non-Small Cell Lung Cancer (NSCLC) Patients With Unresectable Stage III Disease
Brief Title: Safety Study of Tecemotide (L-BLP25) in Non-Small Cell Lung Cancer (NSCLC) Subjects With Unresectable Stage III Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B25-LG-305 / EMR 63325-006
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms
Keywords: Carcinoma, Non-Small-Cell Lung, L-BLP25, Tecemotide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma | interventions — L-BLP25; Single Person; Cyclophosphamide

ARMS (1):
- Tecemotide(L-BLP25)+Cyclophosphomide+best standard of care (Experimental)
  Interventions: Biological: Tecemotide (L-BLP25); Drug: Single low dose cyclophosphamide; Other: Best standard of care (BSC)

INTERVENTIONS:
Biological: Tecemotide (L-BLP25) — After receiving single low-dose cyclophosphamide, subjects will receive 8 consecutive weekly subcutaneous vaccinations with 1000 microgram (mcg) of tecemotide (L-BLP25) at weeks 0, 1, 2, 3, 4, 5, 6 and 7 followed by maintenance vaccinations (1000 mcg of tecemotide [L-BLP25]) at 6-week intervals, commencing at Week 13, until disease progression is documented.
Drug: Single low dose cyclophosphamide — A single intravenous infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide will be administered 3 days prior to tecemotide (L-BLP25), the first vaccine treatment.
Other: Best standard of care (BSC) — The BSC will be provided at the investigator's discretion, and may include but not be limited to psychosocial support, nutritional support and other supportive therapies.

SUMMARY:
The primary objective is to document the safety of tecemotide (L-BLP25) phase III formulation in non-small cell lung cancer (NSCLC) subjects with unresectable Stage III disease. This population includes Stage IIIA NSCLC subjects, a population not studied in former clinical studies with this vaccine. The secondary objective is to document the survival of subjects treated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented unresectable stage III NSCLC. Mediastinal (N2) involvement must be confirmed by biopsy
* Stable disease or clinical response after primary therapy of chemo-radiation treatment for unresectable stage III disease
* Primary therapy should be a minimum of 2 cycles of Platinum-based first-line chemotherapy, given concurrent with thoracic radiation. The combined modality should consist of either:

  * induction (2 cycles) chemotherapy followed by concurrent chemo-radiation therapy; or
  * concurrent chemo-radiation therapy followed by 2 cycles of consolidation chemotherapy; or
  * concurrent chemoradiation therapy alone
* A minimum radiation dose of greater than or equal to (>=) 6,000 centigray (cGy) should be administered. Subjects must have completed the primary therapy at least 4 weeks and no later than 6 months prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to (<=) 1
* Ability to understand and willingness to sign a written informed consent
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Undergone lung cancer specific therapy (including surgery) prior to primary chemo-radiation therapy
* Received immunotherapy/systemic immunosuppressive drugs/investigational systemic drugs within 4 weeks prior to study entry
* Subjects with brain metastases, pleural effusion, unless cytologically confirmed to be non-malignant
* Past or current history of neoplasm other than lung carcinoma, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least 5 years
* Autoimmune disease or immunodeficiency
* Clinically significant hepatic, renal dysfunction or cardiac diseases
* Clinically significant active infection
* Pregnant or lactating, women of childbearing potential, unless using effective contraception as determined by the investigator
* Other protocol defined inclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-04; Primary Completion 2007-09 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany

REFERENCES:
- [Result] Butts C, Murray RN, Smith CJ, Ellis PM, Jasas K, Maksymiuk A, Goss G, Ely G, Beier F, Soulieres D. A multicenter open-label study to assess the safety of a new formulation of BLP25 liposome vaccine in patients with unresectable stage III non-small-cell lung cancer. Clin Lung Cancer. 2010 Nov 1;11(6):391-5. doi: 10.3816/CLC.2010.n.101. PMID 21071331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): April 2005/September 2005. Last participant completed: April 2012; Clinical data cut-off: 17 September 2007. The study was conducted at 8 centers in Canada.
Pre-assignment Details: Enrolled: 22 participants.
Groups:
- Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care: A single intravenous infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide was administered 3 days prior to tecemotide (L-BLP25) first vaccine treatment followed by weekly subcutaneous vaccinations of 1000 microgram (mcg) of tecemotide (L-BLP25) at Week 0, 1, 2, 3, 4, 5, 6, and 7 in the primary treatment phase. Maintenance dose of 1000 mcg of tecemotide (L-BLP25) was administered subcutaneously in the deltoid or triceps region of the upper arms, and the left and right anterolateral aspects of the abdomen at a 6-week intervals, starting at Week 13, until disease progression was documented. The best standard of care (BSC) was provided at the investigator's discretion, and included psychosocial support, nutritional support and other supportive therapies as required.
Period: Overall Study
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care
Started | 22
Completed | 13
Not Completed | 9
Not completed — Ongoing at data cut-off | 9

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) analysis set included all the enrolled participants who received at least 1 dose of trial treatment.
Groups:
- Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care: A single intravenous infusion of 300 mg/m^2 (to a maximum 600 mg) of cyclophosphamide was administered 3 days prior to tecemotide (L-BLP25) first vaccine treatment followed by weekly subcutaneous vaccinations of 1000 mcg of tecemotide (L-BLP25) at Week 0, 1, 2, 3, 4, 5, 6, and 7 in the primary treatment phase. Maintenance dose of 1000 mcg of tecemotide (L-BLP25) was administered subcutaneously in the deltoid or triceps region of the upper arms, and the left and right anterolateral aspects of the abdomen at a 6-week intervals, starting at Week 13, until disease progression was documented. The BSC was provided at the investigator's discretion, and included psychosocial support, nutritional support and other supportive therapies as required.
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs With CALGB-ECTC Grade 3 or 4, TEAEs Leading to Discontinuation, TEAEs Leading to Death, and Injection Site Reactions (ISRs)
Description: TEAEs occurred between the first dose of study drug and up to 42 days after the last dose that were absent before treatment or that worsened relative to pretreatment state. A serious TEAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs with Cancer and Leukemia Group B Extended Clinical Toxicity Criteria (CALGB-ECTC) Grade 3 or 4 were also reported.
Time Frame: Up to data cut-off date (17 September 2007)
Population: Safety analysis set included all the enrolled participants who received at least one dose of the trial treatment.
Measure: Number; unit: participants
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care
Number analyzed (Participants) | 22
participants
  TEAEs | 22
  Serious TEAEs | 4
  TEAEs with CALGB-ECTC Grade 3 or 4 | 13
  TEAEs leading to death | 1
  ISRs | 11

2. Secondary Outcome: Survival Time
Description: Survival time was to be measured from study entry (date of cyclophosphamide administration) to date of death. For subjects alive or lost to follow-up at time of analysis, the time between date of cyclophosphamide administration and date on which the subject was last known alive was to be calculated and used as a censored observation in the analysis.
Time Frame: Up to data cut-off date (17 September 2007)
Population: Safety analysis set included all the enrolled participants who received at least one dose of the trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care
Number analyzed (Participants) | 22
months | NA [17.5 to NA] — The median survival time could not be estimated as there were only eight events reported, still fewer than the 11 events necessary to estimate a median survival time.

3. Secondary Outcome: Progression Free Survival (PFS) Time
Description: PFS was defined as duration from first administration of trial treatment until progressive disease [PD] (radiological or clinical, if radiological progression is not available) or death due to any cause. Participants without event were censored on the date of last tumor assessment. Clinical assessments were performed 4 weekly in primary treatment and 6 weekly in maintenance treatment.
Time Frame: Up to data cut-off date (17 September 2007)
Population: Safety analysis set included all the enrolled participants who received at least one dose of the trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care
Number analyzed (Participants) | 22
months | NA [5.7 to NA] — The PFS could not be estimated as there were only eight events reported, still fewer than the 11 events necessary to estimate a median PFS

ADVERSE EVENTS:
Time Frame: Time from first dose of cyclophosphamide until 42 days following the last vaccination of tecemotide (L-BLP25) or until the data cut-off date (17 September 2007)
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care (N=22)
Coronary artery insufficiency (Cardiac disorders) | 1
Chest pain (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25)+Cyclophosphamide+Best Standard of Care (N=22)
Tachycardia (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 6
Chills (General disorders) | 2
Early satiety (General disorders) | 2
Fatigue (General disorders) | 12
Influenza like illness (General disorders) | 6
Injection site bruising (General disorders) | 5
Injection site erythema (General disorders) | 5
Injection site pain (General disorders) | 3
Pyrexia (General disorders) | 3
Bronchitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 2
Radiation fibrosis - lung (Injury, poisoning and procedural complications) | 2
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2
Weight increased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 8
Hypoaesthesia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 2
Sinus headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study as a whole will be published prior to any individual investigator publications. It is required that copies of all papers, abstracts, articles, etc. that contain study data are to be forward to the Sponsor for review 30 days prior to submission for publication.